CLINICAL TRIAL: NCT04272229
Title: Cognitive Function and Autonomic Regulation in Patients With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fortaleza University (Other)
Responsible Party: Principal Investigator, Mayron F. Oliveira, Clinical Professor, Fortaleza University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 3.741.233
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Cognitive tests will be performed to check if cognition is impaired in patients with migraine compared to healthy control. An R-R ECG recording will be recorded to evaluate the heart rate variability and then the sympathetic nervous system activation. Concentration and attention will be recorded with the MindWave headset during all cognitive tests.
  Interventions: Diagnostic Test: Cognition; Diagnostic Test: Sympathetic Nervous System; Diagnostic Test: Concentratio and Attention
- Migrain Group (Experimental): Cognitive tests will be performed to check if cognition is impaired in patients with migraine compared to healthy control. An R-R ECG recording will be recorded to evaluate the heart rate variability and then the sympathetic nervous system activation. Concentration and attention will be recorded with the MindWave headset during all cognitive tests.
  Interventions: Diagnostic Test: Cognition; Diagnostic Test: Sympathetic Nervous System; Diagnostic Test: Concentratio and Attention

INTERVENTIONS:
Diagnostic Test: Cognition — Cognition tests will be performed with questionnaires, which will be applied to the main investigator. Stroop Color test, digit symbol substitution test, Addenbrooke's cognitive examination 3, mini-mental state examination, Montreal Cognitive Assessment, Trail Making Test A e B and Reaction time test will be performed to check the cognition in all volunteers.
Diagnostic Test: Sympathetic Nervous System — The sympathetic activation will be evaluated by heart rate variability. Volunteers will have their hear rate recorded by a frequencymeter and the R-R interval will be analyzed to ch check the central nervous system activation during all cognitive tests.
Diagnostic Test: Concentratio and Attention — Concentration and attention measures will be recorded with the MindWave headset during all cognitive tests. The EEG will be recorded with the MindWave and then alfa wave will be analized to check the attention and concentration levels.

SUMMARY:
Individuals with migraine have impaired cognitive function and worse autonomic function compared to individuals without migraine. Objective: To evaluate the autonomic function and cognition in young individuals with migraine compared to healthy individuals without migraine. Methods: Cross-sectional study will be carried out at University of Fortaleza with individuals with previous migraines diagnoses and healthy volunteers without migraines. Volunteers of both sexes, aged between 18 and 60 years, clinically diagnosed with migraine or not, who have not undergone any type of drug treatment for at least three months and who accept to participate in the research will be enrolled in the research. Individuals who have comorbidities such as hypertension and Diabetes mellitus (type I and II), respiratory, cardiac and/or chronic vascular diseases, have suffered any significant facial trauma, have a cognitive problem or dysfunction associated with cognition, or have suffered any episode of stroke or transient ischemic attack prior to conducting this research will not be enrolled. Participants will be assessed through cognitive tests, and autonomic function such as Neck Disability Index, Migraine Disability Assessment Questionnaire, Stroop Colo test, digit symbol substitution test, Addenbrooke's cognitive examination, mini-mental state examination, Montreal Cognitive Assessment, Trail Making Test A and B and reaction time test and by MindWave Mobile® devices and Polar V800®.

DETAILED DESCRIPTION:
The sympathetic nervous system is responsible for responding to stressful situations with involuntary actions, which will increase the neuronal activity in order to maintain body homeostasis. Stress is one of the most common causes of migraines. When it occurs for a prolonged period, there will be an over-stimulation of the sympathetic nervous system that will lead to dysautonomia, generating the rapid consumption of the neurotransmitter norepinephrine at the same time that adenosine, dopamine. It is believed that before the headache, the levels of norepinephrine are elevated, causing a vasoconstriction of extracranial vascularization, followed by a vasodilation resulting from the release of the other hormones previously mentioned, thus instituting the painful phase of migraine. Thus, migraine acts on the vascular system through changes in its homeostasis, predisposing the occurrence of future ischemic and/or hemorrhagic episodes to the brain and cardiac levels. The disruption of this system with the multifactorial mechanisms of migraine manifestation can then result in an increased risk of coronary heart disease and other changes in cardiac functioning, acquiring highly harmful potential for the human body. The interest in this study started in view of the numerous uncertainties within the scientific sphere regarding the possible systemic impacts caused by migraines after detailed research on the subject. The same becomes relevant, as it will contribute to the development of knowledge about headaches.

ELIGIBILITY:
Inclusion Criteria:

* Migraine diagnosis

Exclusion Criteria:

* Previous stroke
* Type I or II diabetes
* Heart disease
* vascular diseases
* previous cognition impairment
* mental disorders
* color blindness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Cognition | one week
  Cognitive tests composite will be impaired in the Migraine group compared to healthy subjects. Cognition will be tested by Stroop Color test, digit symbol substitution test, addenbrooke's cognitive examination 3, mini-mental state examination, Montreal Cognitive Assessment, Trail Making Test A e B and reaction time test.
Attention and concentration test | one week
  Concentration and attention will be recorded during the cognition test
Sympathetic activation | one week
  Sympathetic nervous system will be recorded by R-R intervals

CONTACTS AND LOCATIONS:
Overall Officials: Mayron Oliveira, Professor, Principal Investigator — Professor
Locations (1):
- University of Fortaleza, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No